CLINICAL TRIAL: NCT02866149
Title: Analysis of Circulating Tumor Markers in the Blood
Brief Title: Analysis of Circulating Tumor Markers in the Blood (ALCINA)
Acronym: ALCINA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IC 2015-02
Record Dates: First submitted 2016-07-28; First posted 2016-08-15 (Estimated); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Cancer
Keywords: Cancer; circulating tumor biomarkers; circulating tumor DNA; Circulating tumor Cell (CTC)
MeSH Terms: conditions — Neoplasms; Neoplastic Cells, Circulating | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (16):
- Cohort 1 - "Anti checkpoint" (Other): Monitoring of patients with tumours treated by immune therapy.
  Timing of blood sampling:
  * inclusion
  * after #8 weeks on therapy
  * at progression or 6 months from inclusion for patient without progressive disease
  * if toxicity grade 3 or 4, or grade 2 until 1 month.
  Interventions: Biological: Blood sampling
- Cohort 2 - "Oncoscan®" (Other): Monitoring of patients with HER 2+/- breast cancer and correlation with genome-wide copy number, loss of heterozygosity detection, as well as identification of frequently tested somatic mutations (Oncoscan® assays).
  Timing of blood sampling:
  * inclusion
  * after 1 cycle of therapy (weeks 3-4)
  * up to 2 other samples, timepoints decided by the investigator
  Interventions: Biological: Blood sampling
- Cohort 3 - "CirCe-PLA" (Experimental): Feasibility of Proximity-Ligation Assay (PLA) to study membrane proteins dimerisation by on isolated tumour cells in patients with HER2+/- breast cancer (HER 2+/-).
  One tumor sampling.
  Timing of blood sampling:
  * Inclusion
  * up to 3 other samples, timepoints decided by the investigator.
  Interventions: Biological: Blood sampling; Procedure: Tumor sampling
- Cohort 4 - "CDX PDX" (Other): Establishment of xenografts from tumor (PDX) and from Circulating Tumour Cell (CDX) by tumour and blood sampling.
  One tumor sampling.
  Timing of blood sampling:
  * Inclusion
  * up to 3 other samples, timepoints decided by the investigator.
  Interventions: Biological: Blood sampling; Procedure: Tumor sampling
- Cohort 5 - "Post-TP53" (Other): Follow-up of patients previously treated by neoadjuvant chemotherapy for triple negative breast cancer.
  Timing of blood sampling:
  * Inclusion
  * up to 3 other samples, timepoints decided by the investigator.
  Interventions: Biological: Blood sampling
- Cohort 6 - "Palbociclib" (Other): Monitoring of patients treated with palbociclib
  Timing of blood sampling:
  * Inclusion day (2 samples)
  * after #2 weeks of therapy
  * after #4 weeks of therapy
  * at progression.
  Interventions: Biological: Blood sampling
- Cohort 7 - "CTC_PD-L1_Breast" (Other): Detection of PD-L1 in metastatic breast cancer patients
  Timing of blood sampling:
  * Inclusion
  * up to 3 other samples, timepoints decided by the investigator.
  Interventions: Biological: Blood sampling
- Cohort 8 - "CTC_PD-L1_Broncho-Pulmonary" (Other): Detection of PD-L1 in metastatic lung cancer patients
  Timing of blood sampling:
  * Inclusion
  * up to 3 other samples, timepoints decided by the investigator.
  Interventions: Biological: Blood sampling
- Cohort 9 - "NSCLC" (Other): Monitoring of patients with Non-Small Cell lung Cancer treated by immune therapy.
  Blood sampling at 4 timepoints.
  Interventions: Biological: Blood sampling; Procedure: Tumor sampling; Other: Stool sampling
- Cohort 10 - "Palbociclib II" (Other): Monitoring of patient with a metastatic breast cancer treated by palbociclib.
  Timing of blood sampling:
  * Inclusion
  * after #4 weeks of therapy
  * at the first tumoral evaluation (month 3 or 4)
  * at progression.
  Interventions: Biological: Blood sampling
- Cohort 11 - Sarcomas (Other): The cohort includes all patients with bone or soft tissue sarcoma. Timing of blood sampling depending on disease staging.
  Interventions: Biological: Blood sampling
- Cohort 12 - Faslorad (Other): Monitoring of patient with a metastatic breast cancer initiating a treatment by Faslodex-Afinitor.
  Timing of blood sampling:
  * Inclusion
  * after #3-5 weeks of therapy
  * at the first tumoral evaluation (month 2 or 3)
  * at progression.
  Interventions: Biological: Blood sampling
- Cohort 13 - MUm (Other): The cohort concerns patients with uveal melanoma in the 1st systemic line at the metastatic stage (may have had prior adjuvant therapy or surgery/radiofrequency).
  Timing of blood sampling:
  * J1C1
  * J2C1
  * J1C2
  * J1C5 (first tumoral evaluation).
  Interventions: Biological: Blood sampling
- Cohort 14 - CNBC Snipe (Other): This cohort concerns patients with metastatic Non-Small Cell lung Cancer receiving anti-PD-1/PD-L1.
  One tumour sampling.
  Timing of blood sampling:
  * before treatment
  * at W8 of treatment (after radiological examination)
  * at W12 of treatment
  * at progression or 18 months after the beginning of treatment
  Interventions: Biological: Blood sampling; Procedure: Tumor sampling
- Cohort 15 - Breast CLI (Other): This cohort concerns patients with metastatic lobular breast cancer One tumour sampling.
  Timing of blood sampling:
  * At inclusion
  * After biopsy post inclusion (or in 15 days after)
  * after 1 or 2 months of treatment
  * at progression or 18 months after inclusion
  Interventions: Biological: Blood sampling; Procedure: Tumor sampling
- Cohort 16 - Mum immunothérapie (Other): This cohort concerns patients with metastatic uveal melanoma before immunotherapy treatment.
  Timing of blood sampling :
  * at inclusion
  * at cycle 2 or 3 of treatment
  * at the first tumoral evaluation (C5D1)
  * at progression
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — Up to 5 blood samplings can be performed at different time points
Procedure: Tumor sampling — One tumor sampling can be performed, if applicable
  Arms: Cohort 14 - CNBC Snipe; Cohort 15 - Breast CLI; Cohort 3 - "CirCe-PLA"; Cohort 4 - "CDX PDX"; Cohort 9 - "NSCLC"
Other: Stool sampling — Up to 5 blood samplings can be performed at different time points
  Arms: Cohort 9 - "NSCLC"

SUMMARY:
Exploratory study on blood-borne biological markers and their correlation with clinical and pathological characteristics.

DETAILED DESCRIPTION:
Exploratory multi-cohort study including different types of cancer (different organs and/or different histological types).

Each kind of blood-borne biological markers analyses corresponds to a cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with any tumoral disease (proven or suspected), of any type and stage
2. More than18 years old
3. Signed informed consent form

   Additional inclusion criteria if a tumor sample is needed:
4. Tumor considered as accessible by biopsy
5. Normal blood coagulation tests on the last blood analysis

Non-inclusion Criteria:

1. Patient in detention or protected by the law
2. Patient who cannot comply with the study follow up for geographical, social or psychological reasons

   Additional non-inclusion criteria if a tumor sample is needed:
3. Anticoagulant or antiaggregant that cannot be interrupted for the biopsy
4. central-nervous system metastases only (unless a diagnostic or curative surgery is planned before the inclusion in the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 682 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2024-07 (Actual); Study Completion 2024-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of the analysis of different blood-borne tumor biomarkers | 18 months
  Success rate of the tested detection techniques. The success rate of a given detection technique is calculated by the ratio " detection success " / " number of screened patients ".

SECONDARY OUTCOMES:
Correlation with biological and clinical data | 18 months
  Number of biological analysis results correlated to clinical data. Establishment of a proof of concept

CONTACTS AND LOCATIONS:
Overall Officials: François-Clément BIDARD, MD PhD, Study Director — Institut Curie, Paris (FR)
Locations (5):
- France (5):
  - Centre Georges François Leclerc, Dijon
  - Institut du Cancer de Montpellier, Montpellier
  - Institut Curie (Paris hospital), Paris
  - Institut Mutualiste Montsouris, Paris
  - Institut Curie (St Cloud hospital), Saint-Cloud

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).

REFERENCES:
- [Derived] Rodrigues M, Ramtohul T, Rampanou A, Sandoval JL, Houy A, Servois V, Mailly-Giacchetti L, Pierron G, Vincent-Salomon A, Cassoux N, Mariani P, Dutriaux C, Pracht M, Ryckewaert T, Kurtz JE, Roman-Roman S, Piperno-Neumann S, Bidard FC, Stern MH, Renault S. Prospective assessment of circulating tumor DNA in patients with metastatic uveal melanoma treated with tebentafusp. Nat Commun. 2024 Oct 14;15(1):8851. doi: 10.1038/s41467-024-53145-0. PMID 39402032
- [Derived] Eslami-S Z, Cortes-Hernandez LE, Sinoquet L, Gauthier L, Vautrot V, Cayrefourcq L, Avoscan L, Jacot W, Pouderoux S, Viala M, Thomas QD, Lamy PJ, Quantin X, Gobbo J, Alix-Panabieres C. Circulating tumour cells and PD-L1-positive small extracellular vesicles: the liquid biopsy combination for prognostic information in patients with metastatic non-small cell lung cancer. Br J Cancer. 2024 Jan;130(1):63-72. doi: 10.1038/s41416-023-02491-9. Epub 2023 Nov 16. PMID 37973956
- [Derived] Sinoquet L, Jacot W, Gauthier L, Pouderoux S, Viala M, Cayrefourcq L, Quantin X, Alix-Panabieres C. Programmed Cell Death Ligand 1-Expressing Circulating Tumor Cells: A New Prognostic Biomarker in Non-Small Cell Lung Cancer. Clin Chem. 2021 Nov 1;67(11):1503-1512. doi: 10.1093/clinchem/hvab131. PMID 34355741
- [Derived] Darrigues L, Pierga JY, Bernard-Tessier A, Bieche I, Silveira AB, Michel M, Loirat D, Cottu P, Cabel L, Dubot C, Geiss R, Ricci F, Vincent-Salomon A, Proudhon C, Bidard FC. Circulating tumor DNA as a dynamic biomarker of response to palbociclib and fulvestrant in metastatic breast cancer patients. Breast Cancer Res. 2021 Mar 6;23(1):31. doi: 10.1186/s13058-021-01411-0. PMID 33676547
- [Derived] Cabel L, Rosenblum D, Lerebours F, Brain E, Loirat D, Bergqvist M, Cottu P, Donnadieu A, Bethune A, Kiavue N, Rodrigues M, Pierga JY, Tanguy ML, Bidard FC. Plasma thymidine kinase 1 activity and outcome of ER+ HER2- metastatic breast cancer patients treated with palbociclib and endocrine therapy. Breast Cancer Res. 2020 Sep 14;22(1):98. doi: 10.1186/s13058-020-01334-2. PMID 32928264
- [Derived] Jacot W, Mazel M, Mollevi C, Pouderoux S, D'Hondt V, Cayrefourcq L, Bourgier C, Boissiere-Michot F, Berrabah F, Lopez-Crapez E, Bidard FC, Viala M, Maudelonde T, Guiu S, Alix-Panabieres C. Clinical Correlations of Programmed Cell Death Ligand 1 Status in Liquid and Standard Biopsies in Breast Cancer. Clin Chem. 2020 Aug 1;66(8):1093-1101. doi: 10.1093/clinchem/hvaa121. PMID 32712650